CLINICAL TRIAL: NCT05010564
Title: (H-49235) Trivalent Autologous T-Lymphocytes Co-Expressing Three Chimeric Antigen Receptors Targeting CD19, CD20 AND CD22 in Acute B-lineage Leukemia (TRICAR-ALL)
Brief Title: Trivalent CAR-T Cell in Acute B-Lineage Leukemia (TRICAR-ALL)
Acronym: TRICAR-ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Texas Children's Cancer Center (Other)
Responsible Party: Principal Investigator, Bahey Salem MD, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-49235 TRICAR-ALL
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Leukemia, B-Cell
Keywords: Relapsed or refractory B-Cell Leukemia; TRICAR ALL T-Cells; Cyclophosphamide; Fludarabine; immunotherapy; immune effector cell
MeSH Terms: conditions — Leukemia, B-Cell; Recurrence | interventions — Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous TRICAR-ALL T-Cells and lymphodepletion chemotherapy (Experimental): Three dose levels will be evaluated. The TRICAR-ALL T-cells will be administered after lymphodepletion chemotherapy with Cyclophosphamide and fludarabine.
  Interventions: Genetic: Autologous TRICAR-ALL T-cells and lymphodepletion chemotherapy

INTERVENTIONS:
Genetic: Autologous TRICAR-ALL T-cells and lymphodepletion chemotherapy — Three dose levels will be evaluated with the opportunity to dose de-escalate (dose level -1) for toxicity.
  DL-1: 3x10^6 cells/m2
  DL1: 1×10^7 cells/m2
  DL2: 3×10^7 cells/m2
  DL3: 1×10^8 cells/m2
  Lymphodepletion chemotherapy consisting of Fludarabine 30 mg/m2 IV once daily x 4 doses; and Cyclophosphamide 500mg/m2 IV once daily x 2 doses (starting with the first dose of fludarabine)must be completed greater than or equal to 48 hours prior to infusion of CAR-T cells.
  Other Names: Cytoxan; Fludara

SUMMARY:
This is a gene transfer study for patients with a type of blood cancer called Acute Lymphoblastic Leukemia (ALL) that has come back or has not gone away after treatment.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise but have not been strong enough to cure most patients. For example, T lymphocytes can kill cancer cells but there normally are not enough of them to kill all the cancer cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The antibody used in this study targets CD19, CD20 and CD22. This antibody sticks to ALL cells because of a substance on the outside of these cells called CD19, CD20 and/or CD22. For this study, the antibody to CD19, CD20 and CD22 has been changed so that instead of floating free in the blood, it is now joined to the T cells. When T-cells contain an antibody that is joined to them, they are called chimeric antigen receptor- T cells or CAR-T cells.

In the laboratory, we have also found that T cells work better if we also add proteins that stimulate them. One such protein is called 4-1BB. Adding the 4-1BB molecule makes the cells grow better and last longer in the body, giving them a better chance of killing the leukemia cells. In this study we are going to attach the CD19/CD20/CD22 chimeric receptor that has 4-1BB added to the patient's T cells. We will then test how long the cells last.

These T cells, called "TRICAR-ALL" T cells are investigational products not approved by the Food and Drug Administration (FDA) outside the context of a clinical trial.

DETAILED DESCRIPTION:
The TRICAR-ALL T-cells were made in the laboratory by stimulating the patient's blood with growth factors to make the T cells grow. To get the CD19/CD20/CD22 antibody and 4-1BB to attach to the surface of the T cell, we inserted the antibody gene into the T cell. This is done using a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell.

Enrolled patients will be assigned a dose of TRICAR-ALL T-cells. Prior to receiving the TRICAR-ALL T-cells patients will receive two chemotherapy medications, cyclophosphamide (for 2 days) and fludarabine (4 days).

An injection of TRICAR-ALL T-cells will be given into a vein through an IV at the assigned dose. The injection will take from 1 to 20 minutes. Before receiving the infusion of TRICAR-ALL T-cells patients may be pre-medicated with diphenhydramine (Benadryl) and acetaminophen (Tylenol). Patients will be monitored for up to 3 hours after the injection, and will have to remain locally for at least 4 weeks.

If after a 4-week evaluation period, the patient has a complete response, they may proceed to bone marrow transplant, and will be removed from the treatment portion of the study.

Before treatment, patients will undergo a series of tests:

* Physical exam and history
* Blood tests to measure blood cells, serum chemistry, kidney and liver function
* Pregnancy test for female patients who are of childbearing potential
* Measurements of your leukemia tumor cells by bone marrow studies
* Echocardiogram
* Imaging such as PET scans, CT scans or MRIs will be obtained if needed

During and after treatment, patients will receive these standard medical tests:

* History and physical examination: pre-infusion of T cells (pre-Day 0), infusion day (Day 0) and on Days 1, 4, 7, 10, 14, 21, 28, 42, 56 post infusion of T- cells. Subsequently, history will be taken at 3-, 6-, and 12-months post infusion of T-cells, and then yearly for a total of 15 years.
* Blood tests to measure blood cells, serum chemistry, kidney and liver function: pre-infusion of T cells (pre-Day 0), infusion day (Day 0) and on Days 4, 7, 10, 14,21,28,42,56; then at month 3, 6, and 12; then yearly to year 15 (except for blood counts which will be done every 6 months through year 5).
* Viral PCRs: Pre Chemo, infusion day (Day 0), weeks 1-, 2-, 4- and 8; then at month 3, 6, 9 and 12.
* Measurements of your leukemia tumor cells by bone marrow studies at week 4 (+/- 3 days) and week 8 (+/- 3 days) after the infusion and then per standard of care.
* Imaging such as PET scans, CT scans or MRIs will be obtained, if needed, at 4 weeks and again at 8 weeks after T -Cell infusion (+/- 3 days) and then per standard of care.

Blood Draws:

Blood will be taken before the chemotherapy drugs, before T cell infusion, 3-4 hours after the T cell infusion, and on Days 4, 7, 14, 21, 28, 42, 56 ( +/- 3 days) after the infusion; then at month 3, 6, 9, and 12; every 6 months for 4 years, then yearly for a total of 15 years(+/- 2 weeks).

In the event of your death, we will request permission from your next of kin to perform an autopsy to learn more about the effect of this experimental treatment on your cancer.

ELIGIBILITY:
INCLUSION CRITERIA FOR PROCUREMENT:

* Diagnosis of refractory or recurrent B cell Acute Lymphoblastic Leukemia (B-ALL) with expression of CD19, CD20 and/or CD22
* Age between 1 and 25 years.
* Life expectancy of ≥ 8 weeks
* Weight ≥ 10 kg
* Subjects ≥ 18 years of age must have the ability to give informed consent according to applicable regulatory and local institutional requirements. Legal guardian's consent must be obtained for subjects < 18 years of age. Assent will be obtained from pediatric subjects and according to applicable regulatory and local institutional requirements. Adults with cognitive impairment who are unable to consent and those with Down's syndrome are also eligible for this protocol with consent/assent according to applicable regulatory and local institutional requirements.
* The subject must discontinue all anti-cancer agents and, in the opinion of the investigator, has recovered from significant acute toxic effects of: a) Chemotherapy and biologic agents: All chemotherapy and biologic therapy not specifically mentioned below must be discontinued ≥ 7 days prior to collection, with the exception of intrathecal chemotherapy and maintenance chemotherapy being discontinued ≥ 72 hours prior to collection (for the subset of subjects who relapse during maintenance); b) Steroid use: All systemic corticosteroid therapy (unless physiologic replacement dosing of ≤ 12mg/m2/day hydrocortisone or equivalent) must be discontinued ≥ 3 days prior to collection; c) Tyrosine Kinase Inhibitor (TKI) use: All TKIs must be discontinued ≥ 3 days prior to collection; d) Hydroxyurea: must be discontinued ≥ 1 day prior to collection; e) Prior CAR-T cell therapy: must be at least 30 days from most recent CAR-T cell infusion prior to collection; f) Immunotherapy directed at leukemia: No antibodies within three (3) half-lives prior to collection (or within 4 weeks) whichever is shorter. This includes Antithymocyte globulin (ATG) formulations; g) Anti T-cell Antibodies, Alemtuzumab: must be discontinued ≥ 8 weeks prior to collection

EXCLUSION CRITERIA FOR PROCUREMENT:

* Active malignancy other than disease under study
* Presence of active severe infection, defined as: a) positive blood culture within 48 hours of collection, OR; b) known history of active viral infections including infection with HIV, hepatitis B, hepatitis C or HTLV
* Primary immunodeficiency syndrome
* Pregnant or breastfeeding
* Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol

INCLUSION CRITERIA FOR T-CELL THERAPY

* Diagnosis of refractory or recurrent B cell Acute Lymphoblastic Leukemia (B-ALL) with expression of CD19, CD20 and/or CD22 and meeting any of the following conditions:
* B-ALL with no prior history of allo-HCT with one of the following:

  1. Second or subsequent marrow relapse
  2. First marrow relapse if, at the end of re-induction, bone marrow showing ≥ 0.01% blasts by morphology &/or flow cytometry
  3. Primary refractory disease defined by having ≥ 5% blasts in the marrow by morphology and/or minimal residual (MRD) testing after 2 or more separate induction regimens (which may include CD19-targeting therapies)
  4. Subject has an indication for allo-HCT but deemed ineligible (including subjects who have persistent MRD prior to allo-HCT)
  5. CD19(+) or CD19(-) relapse or refractory ALL after infusion of CD19- CAR-T cells or other CD19-targeting immunotherapies. CD20 or CD22 expression is required for CD19(-) B-ALL.

Or

* B-ALL recurrent after allo-HCT defined as having ≥ 0.01% marrow disease
* Available transduced T-cells with ≥ 15% expression of CD19, CD20 or CD22 CAR by flow cytometry.
* Prohibited medications - washout periods (prior to CAR-T cell product infusion): Radiation therapy including TBI and cranial radiation. Local/palliative radiation excluded: ≥ 4 weeks. Cytotoxic chemotherapy: ≥ 2 days. Tyrosine Kinase Inhibitors: ≥ 7 days
* Total Bilirubin: ≤ 3X upper limit of normal (ULN) for age OR conjugated bilirubin ≤ 2mg/dl, except in subjects with Gilbert's syndrome where a total bilirubin level of up to 5.3 mg/dL will be acceptable
* ALT ≤ 5 times upper limit of normal
* Adequate renal function defined as serum creatinine that is ≤ maximum based on age/gender (as indicated below) or Creatinine clearance or GFR (as measured or estimated by Cockcroft Gaultor Schwartz) ≥ 50 mL/min/1.73m2

Maximum Serum Creatinine (mg/dL):

Male and Female: Age 1 to < 2 years: 0.6 Male and Female: Age 2 < 6 years: 0.8 Male and Female: Age 6 to < 10 years: 1.0 Male and Female: Age 10 to < 13 years: 1.2 Male: Age 13 to <16 years 1.5 Female: Age 13 to <16 years 1.4 Male: Age equal to or > 16 years 1.7 Female: Age equal to or > 16 years 1.4

* Pulse oximetry of ≥ 90% on room air
* Left ventricular fractional shortening (LVFS) ≥ 28% confirmed by echocardiogram or left ventricular ejection fraction (LVEF) ≥ 45% confirmed by echocardiogram (MUGA or MRI heart may replace echocardiogram).
* Lansky score of ≥ 50% (age ≥1 and < 16 years) or Karnofsky score of ≥ 50% (age ≥ 16 years). Refer to appendix IV
* Donor lymphocyte infusions (DLI) completed > 6 weeks prior to CAR-T cell infusion
* Subjects of childbearing/fathering potential must agree to use highly effective contraception (see Appendix IIII for acceptable forms of contraception) from the time of initial T cell infusion through 12 months following the last T cell infusion
* Subjects > 18 years of age must have the ability to give informed consent according to applicable regulatory and local institutional requirements. Legal guardian's consent must be obtained for subjects < 18 years of age. Assent will be obtained from pediatric subjects and according to applicable regulatory and local institutional requirements. Adults with cognitive impairment who are unable to consent and those with Down's Syndrome are also eligible for this protocol with consent/assent according to applicable regulatory and local institutional requirements.

Subject willing to participate in long term follow up for up to 15 years.

EXCLUSION CRITERIA FOR T-CELL THERAPY

* Pregnant or lactating
* Presence of any condition that, in the opinion of the PI or designee, would prevent the patient from undergoing protocol-based therapy.
* If history of allogeneic Hematopoietic Cell transplantation (allo-HCT):

  * active GVHD: acute GVHD >/= Grade 2 or chronic GVHD, extensive global severity score, OR
  * actively taking corticosteroids for management of GVHD at a dose of > 0.5 mg/kg/day of prednisone equivalent
  * receiving immunosuppressive therapy for treatment or prevention of GVHD within 4 weeks prior to T-cell infusion.
* Acute symptomatic CNS pathology requiring active medical intervention, including paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder. Subjects with chronic, stable neurological conditions such as non-febrile seizure disorder controlled on anti-epileptic medication and without seizure activity within 3 months may be eligible. Subjects with a history of an isolated seizure episode of ≥ 4 weeks (including methotrexate neurotoxicity) without an underlying epileptic disorder are eligible.

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2040-03-29 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate by CTCAE v5.0 | within 28 days of the TRICAR-ALL T cell infusion.
  Toxicity for all patients will be evaluated using the NCI common toxicity criteria scale, version 5.0 (https://ctep.cancer.gov) with the exception of CRS and neurological toxicities which will be evaluated based on the ASTCT Consensus Guidelines (Lee et al, BBMT 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Bahey Salem, MD, Principal Investigator — Baylor College of Medicine; Nabil Ahmed, MD, Principal Investigator — Baylor College of Medicine; Meenakshi Hegde, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States